CLINICAL TRIAL: NCT05282212
Title: Point of Care, High Resolution and 3-Dimensional Ultrasonography for Diagnosing Peri-Implant Bone Loss
Brief Title: Point of Care, High Resolution and 3-Dimensional Ultrasonography
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Assistant Program Director, Periodontics Graduate Program, University of Michigan
Other Study IDs: HUM00170906
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Bone Loss in Jaw; Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental Implant Surgery: Subjects scheduled for a revision surgery after developing infection after implant surgery
  Interventions: Diagnostic Test: Ultrasound Scan

INTERVENTIONS:
Diagnostic Test: Ultrasound Scan — Within 90 days before the revision surgery, a calibrated examiner will ultrasonically scan the implants. The ultrasound device has been validated for its usability and design on human subjects in our recent clinical study (the University of Michigan Institutional Review Board under the number HUM00139630 and was registered with the National Institutes of Health U.S. National Library of Medicine database for clinical trials (clinicaltrials.gov) under the following identifier: NCT03558282) Coupling will be achieved with commercially available sterilized US gel (Sterile Aquasonic, Fairfield, NJ). The US probe will be mounted on an adjustable arm attached to a fixed stand. The probe is navigated by a calibrated examiner at the implant of interest and then will execute a total ±5 mm linear mesio-distal and coronal-apical translations to create 3D cross-sectional and transverse volumes, respectively and stored as an imageframe series, i.e., a DICOM format cineloop.

SUMMARY:
The overall purpose of this study is to establish an ultrasound technique to aid in oral and dental examination of soft and hard tissues. Ultrasound is currently not used in Dentistry and associated oral examinations and we are exploring its usefulness for clinical practice. This study will investigate the use of ultrasonic imaging for planning and placing dental implants, as well as evaluate the use of ultrasonic imaging for monitoring marginal bone loss around dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* • Have a dental implant infection (bleeding on probing/exudate and probing depths of at least 5 mm) and are or will be scheduled for revision surgery within 90 days of the screening visit.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Unwilling or unable to read and sign informed consent form.
* Pregnancy or unsure of their pregnancy status (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the University of Michigan School of Dentistry who are scheduled for dental implant revision surgery as standard of care in the Graduate Periodontics department.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Dental Implant bone level | Within 90 days before dental surgery
  The difference between ultrasound-determined measurements and intraoperative measurements (optical scanner images as indirect measurements)
Dental implant radicular bone thickness | Within 90 days before dental surgery
  The difference between ultrasound-determined measurements and intraoperative measurements (optical scanner images as indirect measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Hsun-Liang Chan, DDS, MS, Principal Investigator — University of Michigan; Oliver Kripfgans, PhD, Principal Investigator — University of Michigan, Radiology
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Chan HL, Misch K, Wang HL. Dental imaging in implant treatment planning. Implant Dent. 2010 Aug;19(4):288-98. doi: 10.1097/ID.0b013e3181e59ebd. PMID 20683285
- [Background] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Background] Peri-implant mucositis and peri-implantitis: a current understanding of their diagnoses and clinical implications. J Periodontol. 2013 Apr;84(4):436-43. doi: 10.1902/jop.2013.134001. No abstract available. PMID 23537178